CLINICAL TRIAL: NCT00733876
Title: Phase I Clinical Trial, Dose-escalating Intra-aortic Infusion of Allogeneic , Bone Marrow-derived Multipotent Stromal Cells to Prevent and Treat Post-operative Acute Kidney Injury in Patients Who Require On-pump Cardiac Surgery
Brief Title: Allogeneic Multipotent Stromal Cell Treatment for Acute Kidney Injury Following Cardiac Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AlloCure Inc. (Industry)
Collaborators: Intermountain Health Care, Inc. (Other); St Mark's Hospital Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NG-IMC001
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Kidney Tubular Necrosis, Acute
Keywords: Acute Renal Failure Cardiac Surgery Stem Cell
MeSH Terms: conditions — Kidney Tubular Necrosis, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Biological: Multipotent Stromal Cells; Biological: Administration of MSC

INTERVENTIONS:
Biological: Multipotent Stromal Cells — Post-operative administration of MSC
Biological: Administration of MSC — Dose escalation protocol

SUMMARY:
The purpose of this trial is to determine if the administration of allogeneic MSCs at defined doses is safe in patients who are at high risk of developing significant Acute Kidney Injury (AKI) after undergoing on-pump cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Documented ischemic coronary heart and/or valvular heart disease:Acceptable candidate for elective CABG and/or Cardiac Valve Surgery
* Patients at high risk for post-op AKI:Age 18 or older if at high risk for post-op AKI because of underlying Diabetes mellitus (type I or II), CHF, COPD Chronic Kidney Disease (CKD) stage 1-4
* Patients at high risk for post-op AKI :age > 65 or combinations
* Patent femoral artery without aortic aneurysm
* Ability to give informed consent.

Exclusion Criteria:

* Presence of ongoing local or systemic infection
* Younger than 18
* Participation in another clinical trial
* Pregnancy
* Contraindication to general anesthesia
* Prisoner
* Dialysis patient (CKD-6) or patient with CKD-5
* History of malignancy except non-melanoma skin cancer
* Occluded Groin arteries
* Uncontrolled Diabetes mellitus (HbA1c > 10, history of diabetic ketoacidosis or osmolar coma within the last three months)
* Non-healing foot ulcers.
* Clinical evidence of severe peripheral vascular disease (ABI < 0.3)
* Coronary Angiogram < 7 days before surgery
* Inadequate pre-operative time to obtain baseline kidney function data due to urgent/emergent surgery
* Unstable myocardium (evolving myocardial infarction), cardiogenic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Absence of MSC-specific Adverse or Serious Adverse Events | In hospital, monthly x 6, yearly x 3

CONTACTS AND LOCATIONS:
Overall Officials: Christof Westenfelder, MD, Study Director — AlloCure Inc.
Locations (2):
- United States (2):
  - Intermountain Medical Center, Murray, Utah
  - St Mark's Hospital, Salt Lake City, Utah

REFERENCES:
- [Derived] Zhao L, Hu C, Zhang P, Jiang H, Chen J. Preconditioning strategies for improving the survival rate and paracrine ability of mesenchymal stem cells in acute kidney injury. J Cell Mol Med. 2019 Feb;23(2):720-730. doi: 10.1111/jcmm.14035. Epub 2018 Nov 28. PMID 30484934
- [Derived] Westenfelder C, Togel FE. Protective actions of administered mesenchymal stem cells in acute kidney injury: relevance to clinical trials. Kidney Int Suppl (2011). 2011 Sep;1(3):103-106. doi: 10.1038/kisup.2011.24. PMID 25018910
- [Derived] Togel FE, Westenfelder C. Kidney protection and regeneration following acute injury: progress through stem cell therapy. Am J Kidney Dis. 2012 Dec;60(6):1012-22. doi: 10.1053/j.ajkd.2012.08.034. Epub 2012 Oct 2. PMID 23036928